CLINICAL TRIAL: NCT03396276
Title: Houston Emergency Opioid Engagement System (HEROES)
Brief Title: Houston Emergency Opioid Engagement System
Acronym: HEROES
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James Langabeer, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SBMI-17-1021
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Suboxone induction into MAT in the ED (Experimental): Suboxone induction into medication-assisted treatment (MAT) in the emergency department (ED)
  Interventions: Drug: Suboxone; Behavioral: Brief counseling in the ED; Behavioral: Referral to outpatient treatment; Behavioral: Follow-up coaching

INTERVENTIONS:
Drug: Suboxone — 8mg of buprenorphine/2mg of naloxone
Behavioral: Brief counseling in the ED — Patients will receive brief counseling from ED physician prior to discharge about the options for outpatient treatment, as well as opioid dependency.Consented patients will be provided with a pamphlet from the Substance Abuse and Mental Health Services Administration called "Facts About Buprenorphine", as well as an information packet for study contact information for the opioid recovery network providers.
Behavioral: Referral to outpatient treatment — A referral will be made to one of the affiliated MAT clinics.
Behavioral: Follow-up coaching — A designated paramedic with the Houston Fire Department (called the navigator or care coordinator) will work with UTHealth to jointly follow-up on patients both telephonically and in-person. The Houston Fire Department paramedic will provide brief information sharing and assist with coordination in scheduling or registering with MAT clinics or recovery coaching.

SUMMARY:
The Houston Emergency Response Opioid Engagement System (HEROES) is a community-based research program integrating assertive outreach, medication-assisted treatment, behavioral counseling, peer recovery support, and paramedic follow-up in Houston Texas. The objective is to compare differences in engagement and retention in treatment for individuals with opioid use disorder.

DETAILED DESCRIPTION:
The Houston Emergency Response Opioid Engagement System (HEROES) is a non-randomized cohort study based at the University of Texas Health Science Center of Houston. This study seeks to develop an emergency- initiated opioid system of care for individuals with prior opioid overdose and opioid use disorder. The study involves both assertive outreach on individuals who have recent overdoses within the last 72 hours, as well as individuals who are admitted to local hospital emergency departments. The study explores the effect of the combination of assertive outreach, same-day induction into medication-assisted treatment, ongoing maintenance treatment, behavioral counseling, peer recovery support, and paramedic follow-up on patient outcomes. The primary outcome is engagement and retention outpatient treatment. Secondary outcomes include quality of life assessment as well as subsequent relapses and overdoses. The hypothesis is that patients with earlier induction into MAT treatment in the emergency department, who receive routine follow-up, are more likely to engage and be retained in a longer-term treatment program for their addiction.

ELIGIBILITY:
Inclusion Criteria:

* In otherwise good health based on physician assessment and medical history
* Tests positive in urine sample for opioids
* Patients express a willingness to stop opioid use
* Meet Diagnostic and Statistical Manual of Mental Disorders - Text Revision (DSM-IV-TR) criteria for opioid dependence
* Patients must be able to speak English
* Be agreeable to and capable of signing informed consent

Exclusion Criteria:

* Non-English-speaking patients
* Have a known sensitivity to buprenorphine or naloxone
* Be physiologically dependent on alcohol, benzodiazepines or other drugs of abuse that require immediate medical attention. Other substance use diagnoses are not exclusionary.
* Have a medical condition that would, in the opinion of the study physician, make participation medically hazardous, including unstable cardiovascular disease, neurological deficits, trauma, acute hepatitis, stroke, and liver or renal disease)
* Be acutely psychotic, severely depressed, and in need of inpatient treatment, or is an immediate suicide risk
* Be a nursing or pregnant female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient enrollment in outpatient treatment | at the time of enrollment in outpatient treatment
Patient retention in outpatient treatment | 30 days after induction in the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: James R Langabeer, EMT, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing IPD